CLINICAL TRIAL: NCT03839849
Title: Clinical Effectiveness of a Topical Subgingival Application of Injectable Platelet-rich Fibrin as Adjunctive Therapy to Scaling and Root Planing. A Double-blind Split Mouth Randomized Prospective Comparative Controlled Trial
Brief Title: Evaluation of Adjunctive Injectable PRF Therapy Used in Conjunction With Scaling and Root Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Hala Albonni, Dr., Syrian Private University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPU-DN-Perio-1
Record Dates: First submitted 2019-01-27; First posted 2019-02-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Pockets
Keywords: periodontal pockets; injectable platelet-rich fibrin; saline
MeSH Terms: conditions — Periodontal Pocket | interventions — proliferation regulatory factors, human urine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF (Test) (Experimental): injected subgingivally i-PRF after scaling and root planing
  Interventions: Procedure: : i-PRF
- saline (Control) (Active Comparator): injected subgingivally saline after scaling and root planing
  Interventions: Procedure: saline

INTERVENTIONS:
Procedure: : i-PRF — The description of this intervention has been already given before
  Arms: i-PRF (Test)
Procedure: saline — The description of this intervention has been already given before
  Arms: saline (Control)

SUMMARY:
Clinical evaluation of local administration of injectable PRF (injectable platelet-rich fibrin) in periodontal pockets as adjunctive therapy to scaling and root planing. 15 periodontal patients will receive a through traditional mechanical treatment (scaling and root planing). Each patient will receive subgingival i-PRF injected in half mouth and the opposite side will be injected with saline, immediately after the deep scaling session.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy of i-PRF subgingival injection right after scaling and root planing as adjunctive therapy to traditional mechanical therapy. 15 periodontal patients will receive traditional mechanical supra and subgingival scaling and root planing. I-PRF will be applied subgingivally in the deep pockets in a half mouth design. The injected half mouth (study group) for each patient will be allocated randomly. The opposite side will be injected with saline (control group). Clinical parameters will be evaluated: plaque index (PI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL). Clinical measurements will be performed at baseline and at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients are in general good health.
* Patients are from both gender and are adult.
* A sign informed consent from participation and permission to use obtained data for research purposes.
* They have not taken medication known to interfere with periodontal tissue health or healing in the preceding 6 months.
* Presence of bilateral periodontal pockets (≥5 mm) on the minimum of 2 teeth in each side.

Exclusion Criteria:

* Patients less than 18 years' old
* Immunosuppressive systemic diseases (like cancer, AIDS, diabetes…)
* clotting and Hematological disorders
* Medications influence on the gingival and periodontal tissues (like calcium channel blockers, or Long-term steroid use
* The teeth with poor bad filling and poorly fitted restorations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | baseline, 2 months
  measure as the change in distance from the cementoenamel junction to the bottom of the gingival sulcus by using a periodontal probe (UNC 15 "University of North Carolina")
Probing pocket depth (PD) | baseline, 2 months
  measure as the change in distance from the gingival margin GM to the bottom of the gingival sulcus by using a periodontal probe (UNC 15 "University of North Carolina")

SECONDARY OUTCOMES:
full mouth Plaque Index Quigely Hein Index (modified by Turesky et al, 1970) | baseline, 2 months
  0 No plaque
  1. Separate flecks of plaque at the cervical margin of the tooth
  2. A thin continuos band of plaque (up to one mm) at the cervical margin of the tooth
  3. A band of plaque wider than one mm but covering less than one-third of the crown of the tooth
  4. Plaque covering at least one-third but less than two-thirds of the crown of the tooth
  5. Plaque covering two-thirds or more of the crown of the tooth labial/ buccal and lingual surfaces are assessed after using disclosing solution.
  An index for the entire mouth is determined by dividing the total score by the number surfaces examined.
Modified Gingival Index (Trombelli et al. 2004) | baseline, 2 months
  0 = Normal gingiva;
  1. = Mild inflammation - slight change in color and slight edema;
  2. = Moderate inflammation - redness, edema and glazing;
  3. = Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
  will be evaluated visually
Bleeding on probing (BOP) | baseline, 2 months
  All six sites of all teeth are assessed with regard to whether probing elicits bleeding (+) or not (-). The severity of gingivitis is expressed as a percentage.
  - no bleeding upon probing (not recorded)
  + bleeding upon probing
  Calculation:
  BOP= Number of bleeding sites x100/ Number of sites evaluated will be evaluated visually and used a UNC-15 mm "University of North Carolina" periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Hala Albonni, DDS MSc, Principal Investigator — Syrian Private University; Hazem Sawaf, DDS MSc PhD, Study Chair — Syrian Private University
Locations (1):
- Syrian Private University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995
- [Background] Varela HA, Souza JCM, Nascimento RM, Araujo RF Jr, Vasconcelos RC, Cavalcante RS, Guedes PM, Araujo AA. Injectable platelet rich fibrin: cell content, morphological, and protein characterization. Clin Oral Investig. 2019 Mar;23(3):1309-1318. doi: 10.1007/s00784-018-2555-2. Epub 2018 Jul 12. PMID 30003342
- [Background] Wang X, Zhang Y, Choukroun J, Ghanaati S, Miron RJ. Effects of an injectable platelet-rich fibrin on osteoblast behavior and bone tissue formation in comparison to platelet-rich plasma. Platelets. 2018 Jan;29(1):48-55. doi: 10.1080/09537104.2017.1293807. Epub 2017 Mar 29. PMID 28351189
- [Background] Wang X, Zhang Y, Choukroun J, Ghanaati S, Miron RJ. Behavior of Gingival Fibroblasts on Titanium Implant Surfaces in Combination with either Injectable-PRF or PRP. Int J Mol Sci. 2017 Feb 4;18(2):331. doi: 10.3390/ijms18020331. PMID 28165420
- [Background] Kour P, Pudakalkatti PS, Vas AM, Das S, Padmanabhan S. Comparative Evaluation of Antimicrobial Efficacy of Platelet-rich Plasma, Platelet-rich Fibrin, and Injectable Platelet-rich Fibrin on the Standard Strains of Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans. Contemp Clin Dent. 2018 Sep;9(Suppl 2):S325-S330. doi: 10.4103/ccd.ccd_367_18. PMID 30294166